CLINICAL TRIAL: NCT05362643
Title: Effect of Acupuncture on Functional Capacity and Health-Related Quality of Life of Hemodialysis Patients: Randomized Controlled Trial.
Brief Title: Effect of Acupuncture on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Marta Raquel Custódio Correia de Carvalho, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPorto_MCC
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Acupuncture Therapy; Hemodialysis Patients; Quality of Life; Activities of Daily Living
Keywords: Chronic Kidney Disease; Hemodialysis; Acupuncture; Activities of daily living; Health-Related Quality of Life.
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture Group (Experimental): Experimental groups were divided into subgroup A and B and both received a total of 9 acupuncture treatments. However Acupuncture Subgroup A received 3 acupuncture sessions over 3 weeks and Acupuncture Subgroup B received 1 acupuncture session for 9 weeks. The same selection of acupuncture points were applied to both subgroups.
  Interventions: Other: Acupuncture
- Sham Acupuncture Group (Placebo Comparator): Sham Acupuncture groups were also divided into subgroup A and B and both received a total of 9 treatments. Sham Acupuncture subgroup A received 3 sessions over 3 weeks and Sham Acupuncture subgroup B received 1 session for 9 weeks.
  Sham Acupuncture subgroups received acupuncture on non-acupuncture points.
  Interventions: Other: Sham Acupuncture
- Non-Acupuncture Group (No Intervention): Non-acupuncture treatment.

INTERVENTIONS:
Other: Acupuncture — Manual acupuncture on acupoint Tai Xi(KI3), bilateral;Sanyinjiao (SP6), bilateral; Zusanli (ST36), bilateral; Shenmen (HT7) unilateral, in the arm without arteriovenous fistula;Guan Yuan (CV4), unilateral, attempt to achieve De qi sensation. After generating needling sensation, needles were manipulated for one minute, every ten minutes during needle retention (20 minutes), using Sterilized stainless steel needle (0,25x25mm; Tewa, asia-med GmbH).
  Arms: Acupuncture Group
Other: Sham Acupuncture — Manual acupuncture performed as superficial needling (5mm depth) on non-acupuncture points without an attempt to achieve De qi sensation and without stimulation, lasting 20 minutes, using Sterilized stainless steel needle (0,25x25mm; Tewa, asia-med GmbH).
  Arms: Sham Acupuncture Group

SUMMARY:
The proposed randomized controlled trial (RCT) evaluated the effect of acupuncture treatment on the functional capacity (FC) and health-related quality of life (HRQoL) in stage 5 Chronic Kidney Disease (CKD) patients receiving maintenance dialysis. A total of 60 end-stage renal disease (ESRD) patients undergoing hemodialysis (HD) from a dialysis centre (Portugal), were randomly assigned to acupuncture, sham and control group.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) patients undergoing hemodialysis (HD) experience multiple physical and emotional problems, undergo a complex and demanding treatment regimen, face a disruptive chronic disease with a significant decrease in functional capacity and a high impact on their HRQoL. Traditional Chinese Medicine (TCM) has been progressively more accepted as an effective therapeutic approach. The fundamental questions guiding our entire research project were: What is the effect of TCM therapeutic strategies in the improvement of symptoms resulting from renal replacement therapy, in ESRD patients undergoing HD? Does acupuncture have a positive effect on FC and HRQoL of hemodialysis patient? If so, are the results maintained over the long term? And what is the effectiveness of short-term intensive interventions when compared to less frequent and prolonged interventions over time? Is it possible to integrate acupuncture into the dialysis care routine? Based on previous research questions and the complexity of CKD, the objectives of our study were: 1) to assess the effect of acupuncture on FC and HRQoL of ESRD patients undergoing hemodialysis; 2) evaluate the specific effects of acupuncture as compared to sham; 3) evaluate short and long term effects of acupuncture; 4) determine the difference between short-term intensive and ongoing but less-frequent acupuncture treatments; 5) to assess the feasibility of integrating acupuncture on dialysis care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18 years or older, receiving regular hemodialysis (HD) treatment for more than 3 months, 3-times a week session, 4h per session, with medically stable condition.

Exclusion Criteria:

* Patients that refuse to participate in the study, who have a clinical indication that prevents their participation in the study and patients with other comorbidities as poorly controlled malignant hypertension, unstable angina, uncontrolled diabetes mellitus, cerebrovascular failure with recurrent syncope, uncontrolled heart failure, severe mental illness or cognitive impairment will be excluded. Other conditions such as inability to practice physical exercise, have had acupuncture treatment in the past two weeks, known hypersensitivity reaction and/or other side effects after acupuncture treatment, inability to cooperate with the procedures inherent to the application of the procedure, will be also excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Performance on activities of daily living (ADL´s) | Baseline.
  Change in functional capacity (FC) and performance on ADL´s were measured by 6-Minute Walk Test (6MWT).
  The 6MWT is a practical, simple, self-paced walking test that assesses the submaximal level of functional exercise capacity. Changes in the 6 minute walk distance will be used to evaluate the efficacy of therapeutic interventions.
Performance on activities of daily living (ADL´s) | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Change in functional capacity (FC) and performance on ADL´s were measured by 6-Minute Walk Test (6MWT).
  The 6MWT is a practical, simple, self-paced walking test that assesses the submaximal level of functional exercise capacity. Changes in the 6 minute walk distance will be used to evaluate the efficacy of therapeutic interventions.
Performance on activities of daily living (ADL´s) | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Change in functional capacity (FC) and performance on ADL´s were measured by 6-Minute Walk Test (6MWT).
  The 6MWT is a practical, simple, self-paced walking test that assesses the submaximal level of functional exercise capacity. Changes in the 6 minute walk distance will be used to evaluate the efficacy of therapeutic interventions.
Performance on activities of daily living (ADL´s) | Follow up (12 weeks post-treatment).
  Change in functional capacity (FC) and performance on ADL´s were measured by 6-Minute Walk Test (6MWT).
  The 6MWT is a practical, simple, self-paced walking test that assesses the submaximal level of functional exercise capacity. Changes in the 6 minute walk distance will be used to evaluate the efficacy of therapeutic interventions.
Health-Related Quality of Life | Baseline.
  Assessed by Kidney Disease Quality of Life- Short Form (KDQOL-SFTM 1. 3). The KDQOL-SF contains eight generic subscales that assess various aspects of health-related quality of life (HRQOL) and has been widely used in CKD.
Health-Related Quality of Life | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Assessed by Kidney Disease Quality of Life- Short Form (KDQOL-SFTM 1. 3). The KDQOL-SF contains eight generic subscales that assess various aspects of health-related quality of life (HRQOL) and has been widely used in CKD.
Health-Related Quality of Life | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Assessed by Kidney Disease Quality of Life- Short Form (KDQOL-SFTM 1. 3). The KDQOL-SF contains eight generic subscales that assess various aspects of health-related quality of life (HRQOL) and has been widely used in CKD.
Health-Related Quality of Life | Follow up (12 weeks post-treatment).
  Assessed by Kidney Disease Quality of Life- Short Form (KDQOL-SFTM 1. 3). The KDQOL-SF contains eight generic subscales that assess various aspects of health-related quality of life (HRQOL) and has been widely used in CKD.

SECONDARY OUTCOMES:
Lower limbs strength | Baseline.
  Measured by 30 second Sit-to-Stand (STS-30) Test.
Lower limbs strength | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Measured by 30 second Sit-to-Stand (STS-30) Test.
Lower limbs strength | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Measured by 30 second Sit-to-Stand (STS-30) Test.
Lower limbs strength | Follow up (12 weeks post-treatment).
  Measured by 30 second Sit-to-Stand Test.
Handgrip strength | Baseline
  Measured by Hand Grip Strength (HGS) Test, using a digital dynamometer. HGS test is commonly used as an indicator of overall muscle strength.
Handgrip strength | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Measured by Hand Grip Strength (HGS) Test, using a digital dynamometer. HGS test is commonly used as an indicator of overall muscle strength.
Handgrip strength | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Measured by Hand Grip Strength (HGS) Test, using a digital dynamometer. HGS test is commonly used as an indicator of overall muscle strength.
Handgrip strength | Follow up (12 weeks post-treatment).
  Measured by Hand Grip Strength (HGS) Test, using a digital dynamometer. HGS test is commonly used as an indicator of overall muscle strength.

OTHER OUTCOMES:
Demographic and clinical variables | Baseline
  Collected by Sociodemographic and Clinical Data Collection Form.
Pre-intervention questionnaire | Baseline
  Participants who received acupuncture or sham acupuncture (acupuncture or sham acupuncture) answered a questionnaire about their expectations regarding the treatment.
Pos-intervention questionnaire | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Participants who received acupuncture (acupuncture and sham acupuncture groups) answered a questionnaire to assess the degree of discomfort felt in the acupuncture treatment, the concealment of the treatment, the perception of the results and the interference of the acupuncture treatment in the routine of hemodialysis.
Pos-intervention questionnaire | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Participants who received acupuncture (acupuncture and sham acupuncture groups) answered a questionnaire to assess the degree of discomfort felt in the acupuncture treatment, the concealment of the treatment, the perception of the results and the interference of the acupuncture treatment in the routine of hemodialysis.
Blood analytical data | Baseline.
  Blood Tests
Blood analytical data | After Treatment: 3 weeks after baseline assessment (subgroup A).
  Blood Tests
Blood analytical data | After Treatment: 9 weeks after baseline assessment (subgroup B).
  Blood Tests
Blood analytical data | Follow up (12 weeks post-treatment).
  Blood Tests

CONTACTS AND LOCATIONS:
Overall Officials: Marta RC Correia de Carvalho, M.Sc, Principal Investigator — ICBAS School of Medicine and Biomedical Sciences - Oporto University, Portugal
Locations (1):
- Marta Raquel Custódio Correia de Carvalho, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No